CLINICAL TRIAL: NCT04239560
Title: Preventive Effect of Boron-based Gel on Radiation Dermatitis in Patients With Breast Cancer: Phase III Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Preventive Effect of Boron-based Gel on Radiation Dermatitis
Acronym: boron_gel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tabriz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Saeid Safiri, Assistant Professor of Epidemiology, Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TBMZ-Radio-boron gel
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Radiodermatitis
Keywords: Radiodermatitis; Gel; Boron; Radiotherapy; Breast Cancer
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The aim of the study was fully described to the eligible subjects and informed consent was gathered. Afterwards, the patients were assigned into the intervention and placebo groups. In the intervention and placebo groups, subjects received daily a gel containing 3% sodium pentaborate pentahydrate and gel free of any chemical treatment respectively 15 minutes before the radiotherapy session. As the gels were used on the target areas of the patients by the researchers, there was no compliance problem in this study. Afterwards, the study's outcomes were examined at 25th day of treatment for the patients in two groups.
Who Masked: Participant, Care Provider
Masking Description: A gel that has an active ingredient in boron with a gel that does not have a substance and is used as a placebo is completely identical in terms of the shape and size of the container, and the gels themselves do not differ in terms of odor and color, and are completely indistinguishable. (This action was taken by the pharmaceutical company). The important point is that the patient is told that the gel used for the patient may be medication or medication. Clinicians and blind patients will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boron-based Gel (Experimental): During each radiation therapy session, 15 minutes before radiotherapy, 3% sodium pentahydrate panteurate will be used.
  Interventions: Drug: Boron-based Gel (Fibore)
- Radiation Traumatic Dermatitis Treated with Placebo (Placebo Comparator): During each radiotherapy session, 15 minutes before radiotherapy, the gel will be free of any chemical treatments
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Boron-based Gel (Fibore) — During each radiotherapy session, 15 minutes before radiotherapy, the gel used and patients followed up.
  Other Names: Fibore
  Arms: Boron-based Gel
Drug: Placebos — During each radiotherapy session, 15 minutes before radiotherapy, the Placebo gel which be free of any chemical used and patients followed up.
  Other Names: No chemical
  Arms: Radiation Traumatic Dermatitis Treated with Placebo

SUMMARY:
Preventive Effect of Boron-based Gel on Radiation Dermatitis

DETAILED DESCRIPTION:
* Study aim: Radiation dermatitis (RD) is observed in more than 90% of breast cancer patients who receive the radiation therapy (RT). In spite of the high number of studies in this area, there is limited high-quality and comparative research that presents definitive findings suggesting the effectiveness of any single intervention for RD prevention. So, the current phase III clinical trial study was conducted to measure the preventive effects of the aforementioned boron-based gel on different outcomes.
* Design: The parallel design, randomized, double blinded and placebo controlled phase III clinical trial was conducted. One-hundred-eighty-one and seventy-six patients aged 18-75 years were assigned to intervention and placebo groups respectively. Patients in intervention and placebo groups received daily a gel containing 3% sodium pentaborate pentahydrate and gel free of any chemical treatment respectively 15 minutes before the RT session. Dermatitis, erythema, dry desquamation, moist desquamation and necrosis were compared between two groups in terms of percent and number needed to treat.
* Settings and conduct: The female breast cancer patients who admitted to the Shahid Madani Hospital were initially assessed during 2018-2019 and those aged 18-75 years old with no previous history of radiotherapy were invited to the study. Pregnant women, patients with unknown dermatitis and those without any willing to participate in this study were excluded. As there was no similar study to compare our outcome studied, we included 30 patients in the pilot study. Afterwards, the sample size of 16 were calculated for each group based on the erythema to ensure the power of 0.8 and type I error of 0.05. However, we increased the sample size of the study to 181 and 76 subjects in intervention and placebo groups respectively to meet the sample size guidelines for Food and Drug Administration Phase III Clinical Trial Studies, address at least 20% attrition rate during the study, and to enhance the randomization efficiency in balancing the patterns of confounding variables between intervention and placebo groups. As there was no usual treatment for the radiation dermatitis in breast cancer patients, increasing the sample size was not ethically questionable.
* Participants/Inclusion and exclusion criteria:

Inclusion: Patients who are admitted to the study are enrolled in the study and have head and neck cancer in the breast, and are between the ages of 18 and 75 years old and have not received radiotherapy before.

Exclusion: Pregnant women, patients with unknown dermatitis and those without any willing to participate in this study were excluded.

* Intervention groups: The aim of the study was fully described to the eligible subjects and informed consent was gathered. Afterwards, the patients were assigned into the intervention and placebo groups. In the intervention and placebo groups, subjects received daily a gel containing 3% sodium pentaborate pentahydrate and gel free of any chemical treatment respectively 15 minutes before the radiotherapy session. As the gels were used on the target areas of the patients by the researchers, there was no compliance problem in this study. Afterwards, the study's outcomes were examined at 25th day of treatment for the patients in two groups.
* Main outcome variables: Dermatitis and its grades including erythema, dry desquamation, moist desquamation and necrosis were considered as main outcomes in this study based on the Radiation Therapy Oncology Group (RTOG) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to the study are enrolled in the study and have head and neck cancer in the breast, and are between the ages of 18 and 75 years old and have not received radiotherapy before.

Exclusion Criteria:

* Pregnant women, patients with unknown dermatitis and those without any willing to participate in this study were excluded.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Radiation Therapy Oncology Group (RTOG) criteria | The study's outcomes were examined at 25th day of treatment for the patients in two groups
  including erythema, dry desquamation, moist desquamation and necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Farshad SeyedNejad, MD, Principal Investigator — Tabriz University of Medical Sciences
Locations (1):
- Shahid Madani Medical & Training Hospital - Department of Radiotherapy, Tabriz, East Azerbaijan Province, Iran

IPD SHARING:
Plan to Share IPD: Yes
all the data will be available after being published.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after being published
Access Criteria: No limitation